CLINICAL TRIAL: NCT03982030
Title: An Open-label, Pilot Clinical Trial of Dalbavancin for the Treatment of Susceptible Gram-positive Infections Requiring Prolonged Intravenous Antibiotic Therapy
Brief Title: Dalbavancin Outpatient Pilot
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00054355
Record Dates: First submitted 2019-06-10; First posted 2019-06-11 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Gram-Positive Bacterial Infections; Soft Tissue Infections
Keywords: Dalbavacin
MeSH Terms: conditions — Gram-Positive Bacterial Infections; Soft Tissue Infections | interventions — dalbavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dalbavancin (Experimental): Participants with susceptible gram-positive infections requiring prolonged parenteral antibiotic therapy will be treated with dalbavancin.
  Interventions: Drug: Dalbavancin

INTERVENTIONS:
Drug: Dalbavancin — Dalbavancin 1.5g IV at day 0, day 8-10
  Other Names: Dalvance

SUMMARY:
The purpose of this research is to determine if a new antibiotic called dalbavancin will work to treat and cure certain infections while reducing the need for daily antibiotics by vein.

DETAILED DESCRIPTION:
A phase 4, single-center, pilot open-label trial assessing the safety and efficacy of dalbavancin in the outpatient therapy of susceptible gram-positive infections requiring prolonged intravenous therapy.

ELIGIBILITY:
Inclusion

* >=18 years of age
* Provide informed consent
* Agreement to attend required follow-up visits with reasonable transportation plan
* Afebrile for at least 24 hours prior to enrollment
* Expected survival ≥3 months
* If female, non-pregnant and non-lactating; all females of child-bearing potential must have a negative pregnancy test prior to study entry and must agree to use a highly effective method of birth control during the study and for one month thereafter.
* Anticipated hospital discharge within 8 days
* Joint and bone infection:
* Sterile site culture positive for susceptible organism
* Participants with bacteremia and right-sided infective endocarditis (IE):

  * 2 or more blood cultures positive for S. aureus (MSSA or MRSA or Streptococci)
  * Blood cultures negative for 72 hours within 7 days on standard of care antibiotic therapy
  * Definite diagnosis of right sided infective endocarditis by Duke Criteria
  * Echocardiographic assessment (TTE or TEE)
* For patients with opioid use disorder and history of injection opioid use,

  * Injection of opioid substances (IOS) in the last 6 months
  * Fulfill criteria for opioid use disorder

Exclusion

* Polymicrobial infection
* Baseline QTc >500 msec
* Creatinine clearance <30 mL per min
* Immunocompromised from neutropenia, AIDS, malignancy, chemotherapy, or receiving immunosuppressant medication including systemic corticosteroids (intranasal or inhaled corticosteroids acceptable)
* Patients with documented allergies to lipoglycopeptides, vancomycin, or teicoplanin
* Concurrent diseases that, in the Investigator's medical judgment, would interfere with the conduct of the study, confound the interpretation of the study results, or endanger the patient's well-being
* For participants with right-sided IE:
* No mitral or aortic valve involvement on echocardiogram
* Large, mobile vegetations (>10mm)
* Perivalvular abscess
* Presence of an intracardiac device (defibrillator or pacer) or prosthetic valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with resolution of infection | Week 6
  Number of participants with no recurrent signs or symptom of infection

SECONDARY OUTCOMES:
Number of participants with development of breakthrough infection - week 6 | Week 6
  Number of participants with worsening signs or symptoms of primary infection or development of new infection.
Number of participants with development of breakthrough infection - Month 6 | Month 6
  Number of participants with worsening signs or symptoms of primary infection or development of new infection.
Number of participants with hospital readmission - week 6 | Week 6
  Number of participants readmitted for the primary infection under treatment or related complication.
Number of participants with hospital readmission - Month 6 | Month 6
  Number of participants readmitted for the primary infection under treatment or related complication.
Number of participants with need for further surgical intervention - week 6 | Week 6
  Number of participants that need surgical intervention for primary infection prior to end of study participation.
Number of participants with need for further surgical intervention - Month 6 | Month 6
  Number of participants that need surgical intervention for primary infection prior to end of study participation.
Number of adverse events leading to discontinuation of study drug -week 6 | Week 6
Number of adverse events leading to discontinuation of study drug - Month 6 | Month 6
Number of participants loss to follow-up - week 6 | Week 6
  Number of participants that fail to receive second planned dalbavacin dose and attend study visits.
  failure to attend scheduled visits after receiving second dalbavancin dose
Number of participants loss to follow-up - Month 6 | Month 6
  Number of participants that fail to receive second planned dalbavacin dose and attend study visits.
  failure to attend scheduled visits after receiving second dalbavancin dose
Costs of antibiotic therapy | Month 6
  Costs of antibiotic therapy will be measured by combined estimated total costs per participant of inpatient and outpatient antibiotic therapy.
Participant Study Questionnaire week 4 | week 4
  Participant satisfaction will be measured using the 5 point scale (4-strongly agree, 3-agree, 2 neutral, 1-disagree, and 0-strongly disagree). Higher scores denote better outcome.
Participant Study Questionnaire week 24 | Month 6
  Participant satisfaction will be measured using the 5 point scale (4-strongly agree, 3-agree, 2 neutral, 1-disagree, and 0-strongly disagree). Higher scores denote better outcome.
Number of participants with reported overdose | Month 6
Number of participants with new enrollment in addiction treatment | Month 6
Number of participants re-admitted for addiction-related issue | Month 6
Time investment per patient required to follow this model | 6 months
  Time investment per patient will be measured by combined time in minutes spent by study and clinical staff on addiction-related phone calls, paperwork and in-person appointments.

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Morse, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No